CLINICAL TRIAL: NCT01138579
Title: Phase I/II Dose-escalation Study of the Investigational Trifunctional Bispecific Anti-CD20 x Anti-CD3 Antibody FBTA05 in Combination With Donor Lymphocyte Infusion (DLI) in Patients With CD20 Positive Chronic Lymphocytic Leukemia (CLL), Low and High Grade Non-Hodgkin´s Lymphoma (NHL) After Allogeneic Stem Cell Transplantation
Brief Title: Study of the Trifunctional Antibody FBTA05 and Donor Lymphocyte Infusion in B-cell Lymphoma After Allogeneic Stem Cell Transplantation
Acronym: STP-LYM-01
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment delayed, trial medication no loner available
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STP-LYM-01-V01
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2015-12

CONDITIONS: Leukemia; Stem Cell Transplantation
Keywords: FBTA05; CD20; CLL; NHL; DLI; allogeneic transplantation; CD20 positive chronic lymphocytic leukemia (CLL); low and high grade non-Hodgkin´s lymphoma (NHL) after allogeneic stem cell transplantation with active disease
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin | interventions — Bi20 antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: FBTA05

INTERVENTIONS:
Drug: FBTA05

SUMMARY:
This study is an investigator driven, open-label, non-randomized, uncontrolled, dose escalating Phase I/II study evaluating the safety and preliminary efficacy of the trifunctional bispecific antibody FBTA05 in combination with donor lymphocyte infusions (DLI) for treatment of relapsed or refractory disease in CD20 positive either low- or high-grade non-Hodgkin´s lymphoma after allogeneic transplantation

ELIGIBILITY:
Inclusion Criteria:

* Patient´s written informed consent
* ≥ 18 years of age; male and female
* Confirmed CLL, low grade NHL or high grade NHL on standard histological or immunophenotypical criteria described in the WHO classification of lymphoid malignancies
* CD20 positivity (if not already confirmed)
* Adequate haematological, liver and kidney functions
* Platelet count ≥25,000mm³ (=25 x 10^9/l)
* Patients with active disease (relapsed/refractory) that survived at least 60 days after allogeneic transplantation
* Eastern Cooperative Oncology Group (ECOG) performance status <=2 (Appendix IV)
* Negative pregnancy test (no more than 2 days before enrolment) and adequate contraception during the study in women of child bearing potential (pre- menopausal, <2 years post-menopausal or not surgically sterile)

Exclusion Criteria:

* Any anti-CD20 and / or any other anti-T cell directed antibody treatments < 3 months before application of FBTA05
* Positivity for human anti-mouse antibodies (HAMAs)
* History of GvHD ° III or IV, or GvHD requiring steroid therapy with more than 10 mg/day
* Known or suspected hypersensitivity to recombinant, murine or rat proteins
* AST/SGOT greater than 10 x ULN (grade 3, CTCAE)
* Bilirubin greater than 5 x ULN (grade 3, CTCAE)
* Creatinine greater than 3.5 mg/dl (grade 3, CTCAE)
* Acute or uncontrolled chronic infections, viral infections at risk of reactivation (e.g.HCV, HBV, HIV)
* Unable or unwilling to comply fully with the protocol
* Any condition which in the judgement of the Investigator would place the subject at undue risk or interfere with the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08 (Estimated); Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Phase I: Determination of the maximum tolerated dose (MTD)
Phase II: Evaluation of preliminary efficacy of FBTA05 in combination with DLI

CONTACTS AND LOCATIONS:
Locations (1):
- 3. Medizinische Klinik, Klinikum rechts der Isar der TU München, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Buhmann R, Michael S, Juergen H, Horst L, Peschel C, Kolb HJ. Immunotherapy with FBTA05 (Bi20), a trifunctional bispecific anti-CD3 x anti-CD20 antibody and donor lymphocyte infusion (DLI) in relapsed or refractory B-cell lymphoma after allogeneic stem cell transplantation: study protocol of an investigator-driven, open-label, non-randomized, uncontrolled, dose-escalating Phase I/II-trial. J Transl Med. 2013 Jul 2;11:160. doi: 10.1186/1479-5876-11-160. PMID 23815981